CLINICAL TRIAL: NCT02048826
Title: Study of Influence of Timing on Motor Learning
Brief Title: FINGER Robot Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, David Reinkensmeyer, Professor of Anatomy and Neurobiology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS#2008-6432
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Cerebrovascular Accident
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FINGER I (Experimental): Subjects participate in 3 weeks of exercising with the experimental device: FINGER robot with first setting at a minimum of 3 days per week, 1 hour per day with the exercise program
  Interventions: Device: FINGER I; Device: FINGER II
- FINGER II (Experimental): Subjects participate in 3 weeks of exercising with the experimental device: FINGER robot with a second setting at a minimum of 3 days per week, 1 hour per day with the exercise program
  Interventions: Device: FINGER I; Device: FINGER II

INTERVENTIONS:
Device: FINGER I — FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting I
Device: FINGER II — FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting II

SUMMARY:
The purpose of this study is to determine the effectiveness of training hand movement using FINGER robot after stroke. FINGER is a robot that measures finger movements and allows users to play computer games using those movements.

DETAILED DESCRIPTION:
Robotic devices can be used to retrain movement after stroke. However, it is unclear how best to assist in movement. Providing physical assistance may improve the flow of proprioceptive information to the nervous system, which may help a person relearn to move a limb. On the other hand, assisting movement with a robot may cause a person to "slack", not trying as hard during therapy. This study will test the effect of different levels of assistance on recovery of finger function during robot-assisted therapy after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years of age
* Have history of stroke affecting the arm, at least 6 months prior to enrollment
* have arm and/or hand weakness as measured on a standard clinical scale
* do not have active major psychological problems, or problems affecting the stroke-affected arm or hand besides the stroke
* do not have active major brain disease other than the stroke
* have absence of pain in the stroke-affected arm and hand

Exclusion Criteria:

* severe stiffness of the arm or hand as measured on a standard clinical scale
* severe problems speaking or understanding speech as measured on a standard clinical scale
* severe reduced level of consciousness
* severe loss ability to sense movement of your limbs as measured on a standard clinical scale
* currently pregnant
* difficulty in understanding or complying with the instructions given by the researcher
* inability to perform the experimental task that will be studied
* increased pain with movement of the stroke-affected arm or hand

Exclusion criteria that will prevent subjects from participating in the MRI:

* Subjects having any implanted metal such as metallic splinters, metallic surgical clips, prosthetic heart valves, pacemakers, neuro-stimulation devices, orthodontic work that contains ferromagnetic materials,
* Subjects whose occupation or activities may cause accidental lodging of ferromagnetic materials, or that may have imbedded metal fragments from military activities, unless cleared by a screening head CT scan
* Subjects with tattoo(s) presenting metallic or ferromagnetic color ingredients or with facial make-up
* Subjects who have claustrophobia
* Subjects who are currently pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reinkensmeyer, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ingemanson ML, Rowe JR, Chan V, Wolbrecht ET, Reinkensmeyer DJ, Cramer SC. Somatosensory system integrity explains differences in treatment response after stroke. Neurology. 2019 Mar 5;92(10):e1098-e1108. doi: 10.1212/WNL.0000000000007041. Epub 2019 Feb 6. PMID 30728310

RESULTS

PARTICIPANT FLOW:
Groups:
- FINGER I: Subjects participate in 3 weeks of exercising with the experimental device: FINGER robot with first setting at a minimum of 3 days per week, 1 hour per day with the exercise program
  FINGER I: FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting I
  FINGER II: FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting II
  FINGER III: FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting III
- FINGER II: Subjects participate in 3 weeks of exercising with the experimental device: FINGER robot with a second setting at a minimum of 3 days per week, 1 hour per day with the exercise program
  FINGER I: FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting I
  FINGER II: FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting II
  FINGER III: FINGER is a robot that measures finger movements and allows patients to play computer game using those movements. Patients will be exercising with FINGER using setting III
Period: Overall Study
Arm/Group | FINGER I | FINGER II
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FINGER I | FINGER II | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 18
  >=65 years | 3 | 9 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Motor and Strength Outcome Measure Using Box and Block Test Measured in Units of Blocks Placed
Description: The primary endpoint was the change in Box and Blocks score, which measures how many blocks a subject can pick up and place in a box in 60 seconds, from baseline to 1-month post-therapy. The higher the scores, the better arm and hand function indicated.
Time Frame: From baseline to 1-month post therapy
Population: The number of blocks participants able to pick up and place in a box in 60 seconds at one month follow up minus the number of blocks participants able to pick up and place in a box in 60 seconds at baseline.
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | FINGER I | FINGER II
Number analyzed (Participants) | 15 | 15
blocks | 2.3 (3.7) | 2.4 (4.6)

2. Secondary Outcome: Motor and Strength Measure Using Action Research Arm Test Measured as a Score
Description: We compared the change in Action Research Arm Test (ARAT) scores from the baseline evaluation to 1-month post-therapy evaluation. The ARAT is a 57-point scale, 0 being the minimum scoreand 57 being the maximum score, that measures upper extremity function, coordination, and dexterity. The higher scores indicate a better outcome.
Time Frame: From baseline to 1-month post therapy
Population: The ARAT score at one-month post-therapy minus ARAT score at baseline on a 57 point scale.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FINGER I | FINGER II
Number analyzed (Participants) | 15 | 15
scores on a scale | 2.5 (3.7) | 3.5 (4.9)

3. Secondary Outcome: Motor, Strength and Sensory Using Fugl-Meyer Test Measured as a Score
Description: The primary outcome measure was the change in Upper Extremity Fugl-Meyer score on a scale of 0 to 66 at one-month post-therapy. The higher the scores, the better arm and hand function indicated.
Time Frame: From baseline to 1-month post therapy
Population: Fugl-Meyer score at one-month post-therapy minus Fugl-Meyer score at baseline on a 66 point scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FINGER I | FINGER II
Number analyzed (Participants) | 15 | 15
units on a scale | 3.7 (3.3) | 1.8 (1.9)

ADVERSE EVENTS:
Arm/Group | FINGER I | FINGER II
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No